CLINICAL TRIAL: NCT01799122
Title: Randomized Clinical Trial Comparing Mini-Arc Precise Pro and the Trans Vaginal Obturator Tape for Surgical Management of Stress Urinary Incontinence
Brief Title: Trial Comparing Mini-Arc Precise Pro and the Trans Vaginal Obturator Tape for Stress Urinary Incontinence
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Ken Maslow, Assistent Professor, University of Manitoba
Purpose: Treatment
Other Study IDs: B2012:047
Record Dates: First submitted 2013-02-22; First posted 2013-02-26 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Stress Urinary Incontinence; Urethral Sling Surgery
MeSH Terms: conditions — Urinary Incontinence, Stress

ARMS (1):
- Precise sling vs TVT-O sling (Active Comparator)
  Interventions: Device: Mini Arc Precise Pro and Trans vaginal obturator sling (TVT-0)

INTERVENTIONS:
Device: Mini Arc Precise Pro and Trans vaginal obturator sling (TVT-0)

SUMMARY:
Randomized comparison of two surgeries for the treatment of female stress urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* women with stress urinary incontinence with a positive cough test
* patient request surgery for treatment

Exclusion Criteria:

* prodominantely overactive bladder
* previous failed procedure
* MUCP <20 cm H2O
* presence of vaginal prolapse > stage 1
* voiding dysfunction (PVR>100 mL)

Min Age: 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Primary Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Cough test at one year from surgery | One year

SECONDARY OUTCOMES:
Subjective symptoms, QOL questionaires | 1 & 2 years post surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Ken Maslow, Winnipeg, Manitoba, Canada

REFERENCES:
- [Derived] Carter E, Johnson EE, Still M, Al-Assaf AS, Bryant A, Aluko P, Jeffery ST, Nambiar A. Single-incision sling operations for urinary incontinence in women. Cochrane Database Syst Rev. 2023 Oct 27;10(10):CD008709. doi: 10.1002/14651858.CD008709.pub4. PMID 37888839